CLINICAL TRIAL: NCT03719560
Title: Early Systemic Central Nervous System Prophylaxis in Diffuse Large B-cell Lymphoma
Acronym: BrUOG-377
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of funding
Sponsor: Brown University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG-377
Record Dates: First submitted 2018-10-23; First posted 2018-10-25 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Methotrexate; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CNS prophylaxis protocol (Experimental): Patients will receive central nervous system prophylaxis protocol using high-dose methotrexate and cytarabine.
  Interventions: Drug: Methotrexate; Drug: Cytarabine

INTERVENTIONS:
Drug: Methotrexate — Systemic methotrexate
  Other Names: Methotrexate sodium
Drug: Cytarabine — Systemic cytarabine
  Other Names: Cytosar-U

SUMMARY:
Phase 2 single-institution trial of early systemic central nervous system prophylaxis in high-risk diffuse large B-cell lymphoma

DETAILED DESCRIPTION:
This is a prospective phase 2 clinical trial of systemic central nervous system prophylaxis among patients with diffuse large B-cell lymphoma at high risk of central nervous system recurrence. The main objective is to evaluate safety and efficacy of early institution of intensive central nervous system prophylaxis in a high-risk group to minimize the risk of a devastating central nervous system recurrence. Patients receive standard primary immunochemotherapy with an addition of planned central nervous system prophylaxis courses on or around day 15 of cycles 2, 4, and 6. Growth factor support and Pneumocystis jirovecii prophylaxis is required. The primary endpoint of this pilot study is protocol-defined toxicity, whereas efficacy (cumulative incidence of central nervous system recurrence) will be a secondary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* New diagnosis of diffuse large B-cell lymphoma, planned first-line therapy using the standard rituximab- and anthracycline-containing regimens
* No central nervous system involvement on initial staging
* Performance status of 0 or 1 (Eastern Cooperative Oncology Group scale)
* Renal function: creatinine clearance >45 ml/min
* Not pregnant; agreeable to contraception
* Written informed consent
* High risk for central nervous system recurrence as determined by one of the following high-risk features:

  1. high central nervous system International Prognostic Index,
  2. testicular, breast, or uterine involvement,
  3. dual expresser or double/triple-hit status,
  4. HIV positive status, or
  5. Molecularly defined high-risk subtype.

Exclusion Criteria:

* pregancy
* unable to provide informed consent
* significant comorbidity in the investigator's judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion with clinically significant toxicity | 1 year
  Clinically significant toxicity as defined in the protocol

SECONDARY OUTCOMES:
Cumulative incidence of central nervous system recurrence | 2 years
  Cumulative incidence of central nervous system recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Adam J Olszewski, MD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Roxanne Wood, Providence, Rhode Island, United States